CLINICAL TRIAL: NCT02549469
Title: A Pilot Four-Way Crossover Bioequivalence Trial of Sustained Release Forms of Naproxen Versus Aleve Tablets in Healthy Adult Subjects in a Fasted State
Brief Title: Bioequivalence of Single Dose Extended Release Naproxen Sodium (660 mg) Tablet Versus Naproxen Sodium (220 mg) Tablet Three Times Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12656
Record Dates: First submitted 2015-08-17; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Naproxen sodium extended release 660 mg, 20% HPMC (Experimental): Bioequivalence in healthy adult subjects in a fasted state relative to the established commercial Aleve (Naproxen sodium) 220 mg tablet
  Interventions: Drug: Naproxen Sodium ER (BAY117031), 20% HPMC
- Naproxen sodium extended release 660 mg, 30% HPMC (Experimental): Bioequivalence in healthy adult subjects in a fasted state relative to the established commercial Aleve 220 mg tablet
  Interventions: Drug: Naproxen Sodium ER (BAY117031), 30% HPMC
- Naproxen sodium extended release 660 mg, 40% HPMC (Experimental): Bioequivalence in healthy adult subjects in a fasted state relative to the established commercial Aleve 220 mg tablet
  Interventions: Drug: Naproxen Sodium ER (BAY117031), 40% HPMC
- Naproxen sodium 220 mg (Active Comparator): Bioequivalence in healthy adult subjects in a fasted state
  Interventions: Drug: Aleve (Naproxen Sodium, BAY117031)

INTERVENTIONS:
Drug: Naproxen Sodium ER (BAY117031), 20% HPMC — 1 tablet 660 mg administered orally once daily
  Arms: Naproxen sodium extended release 660 mg, 20% HPMC
Drug: Naproxen Sodium ER (BAY117031), 30% HPMC — 1 tablet 660 mg administered orally once daily
  Arms: Naproxen sodium extended release 660 mg, 30% HPMC
Drug: Naproxen Sodium ER (BAY117031), 40% HPMC — 1 tablet 660 mg administered orally once daily
  Arms: Naproxen sodium extended release 660 mg, 40% HPMC
Drug: Aleve (Naproxen Sodium, BAY117031) — 1 tablet 220 mg administered orally three times daily
  Arms: Naproxen sodium 220 mg

SUMMARY:
Bioequivalence trial in healthy adult subjects to determine the bioavailability of 3 different sustained release formulations of naproxen 660 mg relative to the established commercial Aleve 220 mg tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory male and female subjects 18 to 55 years of age, inclusive
* Body Mass Index (BMI) of approximately 18.0 to 30.0 kg/m2, and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal limits or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, intramuscular injection or double-barrier and have a negative pregnancy test at Screening and on Day 0 of each treatment period. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy.
* Provide a personally signed and dated informed consent prior to inclusion in the trial indicating that the subject has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), naproxen sodium, or acetaminophen, and similar pharmacological agents or components of the products
* History of gastrointestinal bleeding or perforation, including bleeding related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding).
* Have taken ASA, ASA-containing products, acetaminophen (acetyl-para-amino-phenol or APAP) or any other NSAID (OTC or prescription) 7 days prior to dosing or during the treatment period, other than study treatment
* Loss of blood in excess of 500 mL within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis, or injury)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Positive alcohol or drug screen at Screening or on Day 0 of Treatment Periods 1 or 2
* Females who are pregnant or lactating
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product (eg, nicotine patch, nicotine gum).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum plasma concentration) for naproxen sodium | Days 0, 1, 2, and 3
AUC0-24 (partial area under the curve ) for naproxen sodium | Days 0, 1, 2, and 3
AUC0-t (areas under the curve ) for naproxen sodium | Days 0, 1, 2, and 3
AUC0-∞ (area under the curve) for naproxen sodium | Days 0, 1, 2, and 3
Tmax (The first time point where Cmax is reached) for naproxen sodium | Days 0, 1, 2, and 3
AUC0-8 (partial area under the curve) for naproxen sodium | Days 0, 1, 2, and 3
AUC8-16 (partial area under the curve ) for naproxen sodium | Days 0, 1, 2, and 3
AUC16-24 (partial area under the curve) for naproxen sodium | Days 0, 1, 2, and 3
λz (terminal elimination rate constant) | Days 0, 1, 2, and 3
t1/2 (terminal half life) | Days 0, 1, 2, and 3

SECONDARY OUTCOMES:
Adverse events (AEs) collection | up to 50 days
Serious adverse events (SAEs) collection | up to 50 days
Vital signs: sitting blood pressure | up to 50 days
Vital signs: repiratory rate | up to 50 days
Vital signs : pulse rate | up to 50 days
Clinical Laboratory data | up to 50 days
  Blood and urine samples were collected according to standard medical guidelines at the Screening Visit. In addition, hematology and chemistry were obtained at the end of the study (EOS).
Physical examination findings | up to 50 days
  Brief physical examination, including height, weight and BMI, was performed at the Screening Visit and at EOS

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer